CLINICAL TRIAL: NCT00265213
Title: How Breast Conservative Surgery (BCS) Affects Women's Daily Activities On Post-Operation 2 Days?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Other Study IDs: KMUH-IRB-940194
Record Dates: First submitted 2005-12-12; First posted 2005-12-14 (Estimated); Last update posted 2008-02-27 (Estimated); Status verified 2005-12

CONDITIONS: Breast Cancer
Keywords: breast conservative surgery; shoulder functional outcome questionnaire; disability questionnaire
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
we revise 8 disability items from SPADI into Chinese to develop a simple self-completion questionnaire for the assessment of restriction in daily activities resulting from breast conservative surgery.

The purpose of this study was to validate the score obtained from this questionnaire by testing restriction of shoulder active flexion and abduction on examination at post BCS 2 days correlates with disability score.

DETAILED DESCRIPTION:
Breast-conserving therapy (BCT) is a breast cancer treatment using breast conservative surgery(BCS) with lymph node dissection and with or without following by radiotherapy(RT). (Morrow,2004). Results of BCTs demonstrate high rates of local tumor control with satisfactory cosmetic results. (Morrow,2004) Nowadays, the local treatment of breast cancer has slowly accepted from radical mastectomy with lymph node dissection to (BCT) in the last 100 years. (Morrow,2004) After surgical intervention for breast cancer carcinoma, the most frequent morbilities are lymphedema of the unilateral upper extremity and shoulder dysfunction. (Wingate L,1985; Grube, 2004)From the perspective of the Institute of Medicine's(IOM), the outcome measures shifts from the impairment-based measures to functional limitation measures. (Jette AM,1995) Base on the third element in Donabedian's framework of quality of physical therapy care, the determination of outcomes in terms of death, morbidity, disability, or quality of life. (Jette AM,1995)Although shoulder active range-of-motion exercises could start at the day right after any type or level of lymph node dissections for breast cancer patients, (Staradub VL, 2004;Wingate L,1985) in my literature review results, no functional evaluation questionnaires that was sensitive enough to detect the disabilities resulting from lymph node dissections at post BCS 2 days. So we revise 8 disability items from SPADI into Chinese to develop a simple self-completion questionnaire for the assessment of restriction in daily activities resulting from breast conservative surgery.

The purpose of this study was to validate the score obtained from this questionnaire by testing restriction of shoulder active flexion and abduction on examination at post BCS 2 days correlates with disability score.

ELIGIBILITY:
Inclusion Criteria:

* post breast conservative surgery 2 days
* with lymph node dissection

Exclusion Criteria:

* total SPADI score is not zero

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-05; Study Completion 2006-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ching Chun Lin, PT,CAS, Principal Investigator — Rehabilitation department, Kaoshing Medical University Chung-Ho Memorial Hospital
Locations (1):
- Rehabilitation department,Kaoshing Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan